CLINICAL TRIAL: NCT01405365
Title: The Impact of Obesity on Nonsurgical Periodontal Treatment of Destructive Periodontal Diseases
Brief Title: The Impact of Obesity on Nonsurgical Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Augusta University (Other)
Responsible Party: Cassiano K. Rosing, Faculdade de Odontologia, Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNPq-402335/2008-2
Record Dates: First submitted 2010-08-23; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2010-08

CONDITIONS: Periodontitis; Periodontal Diseases; Obesity
Keywords: Periodontitis; Periodontal diseases; Obesity; Metronidazole; Prognosis; Probing depth; Periodontal attachment loss
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Obesity; Periodontal Attachment Loss | interventions — Metronidazole; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole (Experimental)
  Interventions: Drug: Metronidazole; Procedure: Scaling and root planning
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Procedure: Scaling and root planning

INTERVENTIONS:
Drug: Metronidazole — Metronidazole 400mg TID for 10 days
  Other Names: Flagyl
  Arms: Metronidazole
Drug: Placebo — Placebo pill TID for 10 days
  Other Names: Inactive Substance; Inactive Drug
  Arms: Placebo
Procedure: Scaling and root planning — Scaling and root planning performed with curettes and ultrasonic scalers under local anesthesia
  Other Names: Nonsurgical periodontal therapy

SUMMARY:
The purpose of this study is to investigate the effect that obesity may have on the nonsurgical treatment (with and without the adjunct use of metronidazole) of destructive periodontal diseases (chronic periodontitis).

DETAILED DESCRIPTION:
Normal weight (BMI 18.5-24.9 kg/m2) and obese (BMI >30 kg/m2) women will be randomly assigned to two nonsurgical periodontal treatments:

1. scaling and root planing + placebo
2. scaling and root planing + metronidazole

ELIGIBILITY:
Inclusion Criteria:

* Normal weight or obese (according to BMI)
* nonsmokers or former smokers (3 or more years)
* no systemic diseases that may affect periodontal treatment (diabetes, osteoporosis, steroid use)
* have 10 teeth present
* have at least 2 teeth with probing depth 6+mm and attachment loss 4+mm

Exclusion Criteria:

* Pregnancy
* Development of diabetes or other conditions that may impair periodontal healing

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Probing depth | 12 months
  Defined as the distance from the free gingival margin to the bottom of the pocket/sulcus.

SECONDARY OUTCOMES:
Attachment level | 12 months
  Defined as the distance from the CEJ to the bottom of the pocket/sulcus.

CONTACTS AND LOCATIONS:
Overall Officials: Cassiano K Rosing, DDS, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Cristiano Susin, DDS, PhD, Principal Investigator — Medical College of Georgia School of Dentistry
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil